CLINICAL TRIAL: NCT01299285
Title: Disposition of 14C-LY3009104 Following Oral Administration in Healthy Human Male Subjects
Brief Title: Disposition of 14C-LY3009104 Following Oral Administration in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14010; I4V-MC-JADG (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
Keywords: Absorption; Distribution; Metabolism; Excretion; Mass balance; Metabolic profile; Radiolabeled study; 14C
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY3009104 (Experimental): Single 10-milligram (mg) oral dose containing 100 microcuries of 14C-labeled LY3009104
  Interventions: Drug: LY3009104

INTERVENTIONS:
Drug: LY3009104 — Administered orally
  Other Names: Baricitinib

SUMMARY:
This is a single dose study of radiolabeled [14C]-LY3009104 in healthy male volunteers to study the absorption, distribution, metabolism, and elimination of LY3009104. This study requires minimum of 7 days and maximum of 22 days stay. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males, as determined by medical history and physical examination
* Will either be sterile or, if sexually active, agree to use a reliable method of birth control from check-in until 3 months after the end of the study
* Body mass index (BMI) between 19 and 30 kilogram/square meter (kg/m²)
* Experience on average 1 to 2 bowel movements per day
* Clinical laboratory test results within the normal reference range for the clinical research unit (CRU) or, results with acceptable deviations which are judged to be not clinically significant by the investigator
* Normal blood pressure and heart rate (sitting) as determined by the investigator
* Venous access sufficient to allow blood sampling
* Are reliable and willing to make themselves available for the duration of the study, and are willing to abide by the CRU policies and procedures, and study restrictions
* Have given written informed consent approved by Lilly and the Institutional Review Board (IRB) governing the CRU

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued, a clinical trial involving an investigational product or are concurrently enrolled in any other type of medical research judged not to be scientifically, or medically compatible with this study
* Have known allergies to LY3009104, related compounds, or any components of the formulation
* Have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY3009104
* History or presence of an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, is clinically significant
* Current or recent history (<30 days prior to Screening and/or <45 days prior to Check-in) of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* An Absolute Neutrophil Count (ANC) less than 2000 cells/microliter. For abnormal values a single repeat will be allowed
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Show evidence of significant active neuropsychiatric disease and in particular evidence of significant medical or psychiatric illness within the past 12 months
* Have known substance dependence or abuse within 6 months prior to the study (according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM-IV] diagnosis), or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Evidence hepatitis B (active or surface antigen positive [HBsAg+]) or hepatitis B core antibody positive, hepatitis B surface antibody negative (HBcAb+, HBsAb-)
* Use of prescription medication; over-the-counter medication; or herbal preparations containing St. John's Wort, kava, garlic, ginger, gingko biloba, or guarana within 14 days prior to admission
* Consumption of grapefruit or grapefruit-containing foods or juices within 7 days prior to dosing or at any time during the study
* Have an average weekly alcohol intake that exceeds 15 units per week, or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 oz or 360 milliliter (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any subjects unwilling to adhere to study caffeine restrictions (no caffeine 48 hours prior to admission until the end of study
* Use of tobacco or nicotine-replacement products within the 6 months prior to study entry or at any time during the study
* Have donated blood of more than 500 mL within the last month
* Have participated in a 14C-study within the last 6 months prior to Check-in for this study. The total exposure from this study and the previous study must be within the Code of Federal Regulations (CFR) recommended levels considered safe (per 21 CFR 361.1), for example less than 5,000 millirem (mrem)/year whole body annual exposure
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559, Mon - Fri, 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri, 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3009104 (Baricitinib): Single 10-milligram (mg) oral dose containing 100 microcuries of 14C-labeled LY3009104
Period: Overall Study
Arm/Group | LY3009104 (Baricitinib)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- LY3009104: Single 10-mg oral dose containing 100 microcuries of 14C-labeled LY3009104
Arm/Group | LY3009104
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  White | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Total Radioactive Dose Administered Excreted From Urine and Feces
Time Frame: Baseline up to 120 hours
Population: Participants who took study drug.
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Arm/Group | LY3009104
Number analyzed (Participants) | 6
percentage of total radioactivity
  Urine | 75.2 (6.74)
  Feces | 19.9 (4.92)

2. Secondary Outcome: Plasma Pharmacokinetics: LY3009104 Area Under the Concentration-Time Curve From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Baseline up to 48 hours
Population: Participants who took study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomoles/liter(h*nmol/L)
Arm/Group | LY3009104
Number analyzed (Participants) | 6
hour*nanomoles/liter(h*nmol/L) | 1570 (28)

3. Secondary Outcome: Plasma Pharmacokinetics: Radioactivity Area Under the Concentration-Time Curve From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Baseline up to 48 hours
Population: Participants who took study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole-equivalents/kilogram
Arm/Group | LY3009104
Number analyzed (Participants) | 6
hour*nanomole-equivalents/kilogram | 1530 (31)

4. Secondary Outcome: Plasma Pharmacokinetics: Maximum Observed LY3009104 Concentration (Cmax)
Time Frame: Baseline up to 48 hours
Population: Participants who took study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/liter (nmol/L)
Arm/Group | LY3009104
Number analyzed (Participants) | 6
nanomoles/liter (nmol/L) | 227 (36)

5. Secondary Outcome: Plasma Pharmacokinetics: Maximum Observed Radioactivity Concentration (Cmax)
Time Frame: Baseline up to 48 hours
Population: Participants who took study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole-equivalents/milliliter
Arm/Group | LY3009104
Number analyzed (Participants) | 6
nanomole-equivalents/milliliter | 231 (35)

6. Secondary Outcome: Plasma Pharmacokinetics: LY3009104 and Radioactivity Time to Maximum Observed Concentration (Tmax)
Time Frame: Baseline up to 48 hours
Population: Participants who took study drug.
Measure: Median (Full Range); unit: hour
Arm/Group | LY3009104
Number analyzed (Participants) | 6
hour
  LY3009104 | 1.00 [1.00 to 2.00]
  Radioactivity | 1.00 [1.00 to 2.00]

7. Secondary Outcome: Percentage of Dose of LY3009104 and LY3009104 Metabolites in Urine
Description: Percentages of LY3009104 (parent) and LY3009104 metabolites that were excreted in the urine are reported. Only those metabolites that were detectable in the urine are included in the report.
Time Frame: Baseline up to 48 hours
Population: Participants who took study drug.
Measure: Number; unit: percentage of dose
Arm/Group | LY3009104
Number analyzed (Participants) | 6
percentage of dose
  LY3009104 | 68.5
  Metabolite M3 | 0.9
  Metabolite M10 | 1.0
  Metabolite M22 | 3.2

8. Secondary Outcome: Percentage of Dose of LY3009104 and LY3009104 Metabolites in Feces
Description: Percentages of LY3009104 (parent) and LY3009104 metabolites that were excreted in the feces are reported. Only those metabolites that were detectable in the feces are included in the report.
Time Frame: Baseline up to 72 hours
Population: Participants who took study drug.
Measure: Number; unit: percentage of dose
Arm/Group | LY3009104
Number analyzed (Participants) | 6
percentage of dose
  LY3009104 | 14.8
  Metabolite M12 | 0.9

9. Secondary Outcome: Percentage of Total Radioactivity of LY3009104 and LY3009104 Metabolites in Plasma
Time Frame: Baseline up to 24 hours
Population: Participants who took study drug.
Measure: Number; unit: percentage of total radioactivity
Groups:
- LY3009104: The percentage of total radioactivity of LY3009104 (parent) in the plasma after receiving a single 10-mg oral dose containing 100 microcuries of 14C-labeled LY3009104
- LY3009104 Metabolites: The percentage of total radioactivity of all LY3009104 metabolites in the plasma after receiving a single 10-mg oral dose containing 100 microcuries of 14C-labeled LY3009104
Arm/Group | LY3009104 | LY3009104 Metabolites
Number analyzed (Participants) | 6 | 6
percentage of total radioactivity
  1 hour | 92.3 | 0
  2 hour | 94.5 | 0
  4 hour | 97.0 | 0
  8 hour | 91.2 | 0
  24 hour | 0 | 0

ADVERSE EVENTS:
Arm/Group | LY3009104
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3009104 (N=6)
Ocular hyperaemia (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days